CLINICAL TRIAL: NCT00519103
Title: Resistance Exercise Reduces the Expression of Inflammation and Fibrosis Associated Genes in Autoimmune Myositis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lundberg-1
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: Myositis; Exercise
Keywords: microarray; Inflammtion; fibrosis
MeSH Terms: conditions — Myositis; Motor Activity; Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Active resistive excercise for 7 weeks
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise

SUMMARY:
The aim of this study was to investigate the effects of physical exercise on gene expression in muscle biopsies from patients with chronic polymyositis or dermatomyositis

DETAILED DESCRIPTION:
Eight patients with polymyositis or dermatomyositis according to the Bohan and Peter criteria and who had all participated in a resistive exercise trial at Karolinska University Hospital, Stockholm, Sweden, were included in this study. Patients were included if they had a disease duration more than 12 months and they had to have a stable, low disease activity and medication for three months before enrollment in the study. Patients with inclusion body myositis were excluded as well as patients with co morbidities that contradicted vigorous exercise (severe osteoporosis with multiple fractures, malignant disease severe lung disease) or if they were physically active more than once a week. The median disease duration at time of study start was 4.5 years (range 2,7-29 year). All patients had been treated with glucocorticoids and other immunosuppressive therapies with some improvement of muscle function but with persisting muscle impairment. At time of study seven patients were still on immunosuppressive treatment, five were taking prednisone with a median dosage of 2.5 mg/day (range 0-6.25 mg/d). Six patients were treated with azathioprine, one in combination with cyclosporine A, one patient was treated with methotrexate and one with IVIG 2g/kg body weight every three months

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they had a disease duration more than 12 months and they had to have a stable, low disease activity and medication for three months before enrollment in the study

Exclusion Criteria:

* Patients with inclusion body myositis were excluded as well as patients with co morbidities that contradicted vigorous exercise (severe osteoporosis with multiple fractures, malignant disease severe lung disease) or if they were physically active more than once a week.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-12; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
effects of physical exercise muscle strength and function in patients with chronic polymyositis or dermatomyositis | 7weeks

SECONDARY OUTCOMES:
effects of exercise on gene expression and corresponding protein expression in muscle tissue and on signs of inflammation in peripheral blood | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid E Lundberg, MD, PhD, Principal Investigator — Rheumatology Unit, Department of Medicine, in Solna, Karolinska Institutet
Locations (1):
- Rheumatology unit, Karolinska Unirversity hospital, Stockholm, Sweden